CLINICAL TRIAL: NCT00663013
Title: Virtual Reality for Burn Wound Care Pain Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: R. W Yurt, MD,FACS, NewYork-Presbyterian Hospital-Weill Cornell Medical College
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0701008961
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2011-01

CONDITIONS: Pain; Anxiety
Keywords: burn; pain; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders; Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): The first treatment session will involve 5-7 minutes of burn wound care while distracted by VR, and 5-7 minutes of burn wound care without the distraction of VR. The second session of burn wound care (performed within the next 3 days) will involve 5-7 minutes of burn wound care without the distraction of VR, and 5-7 minutes of burn wound care with the distraction of VR. The treatment order will be randomized.
  Interventions: Other: Virtual Reality
- 2 (Active Comparator): The first treatment session will involve 5-7 minutes of burn wound care while distracted by VR, and 5-7 minutes of burn wound care without the distraction of VR. The second session of burn wound care (performed within the next 3 days) will involve 5-7 minutes of burn wound care without the distraction of VR, and 5-7 minutes of burn wound care with the distraction of VR. The treatment order will be randomized.
  Interventions: Other: Virtual Reality

INTERVENTIONS:
Other: Virtual Reality — Virtual reality (VR) gives patients an illusion of going into the 3-D computer generated environment/virtual world. During VR, the subject wears a head-mounted virtual reality helmet that positions two goggle-sized miniature LCD computer screens close to the subject's eyes. Position tracking devices keep the computer informed of changes in the patient's head location. An electro-magnetic head orientation device feeds the x, y, z coordinates of the patient's head to the computer, which can quickly change what the patient sees in virtual reality accordingly. The scenery in VR changes as the patient moves her head orientation (e.g., virtual objects in front of the patient in VR get closer as the patient, wearing the VR helmet, leans forward in the real world).
  Other Names: SnowWorld Multigen-Paradigm Inc, SimWright Inc

SUMMARY:
The investigators propose to study the effects of virtual reality (VR) on patients' pain perception during burn wound care. Such variables include psychiatric diagnosis and standard pain coping (i.e. pain catastophizer vs. non-pain catastrophizer).Aims: The investigators intend to evaluate the use of virtual reality in pain distraction for burn patients undergoing burn wound care. To that end our aims are: 1) To determine if pain perception will be less during the portion of the procedure in which the patient is immersed in the VR session in comparison to the portion of wound care which will occur without VR immersion. 2) To determine if anticipatory anxiety will be less for the portion of wound care that includes the virtual reality in comparison to the portion without virtual reality. 3) To determine if current psychiatric diagnosis, especially acute stress disorder and depression, is related to higher pain perception and greater decrease in pain with the virtual reality distraction. 4) To determine if being a "pain catastrophizer" is related to higher pain perception and greater benefits from the

ELIGIBILITY:
Inclusion Criteria:

* Age 12-100years
* Minimum burn wound size of 2% total body surface area (TBSA) excluding head and dominant hand
* Be able to sit upright independently in bed
* Minimum pain rating of 4/10 on a Visual Analog Scale (only using the most painful extremity).
* Able to consent to the study

Exclusion Criteria:

* Known history of motion sickness
* Seizures
* Migraines
* Current psychosis, dementia, or delirium
* Current blindness and/or deafness that significantly affects their ability to experience the VR

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
pain perception | immediate
anticipatory anxiety | immediate
current psychiatric diagnosis, is related to pain | immediate
"pain catastrophizing" is related to higher pain perception and greater benefits from the VR | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Roger W Yurt, MD FACS, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital, WRH Burn Center, New York, New York, United States